CLINICAL TRIAL: NCT06026371
Title: Fecal Microbiota Transplantation to Prevent Acute Graft-Versus-Host Disease After Allogeneic Hematopoietic Cell Transplantation
Brief Title: Fecal Microbiota Transplantation for the Prevention of Acute Graft Versus Host Disease in Adults Undergoing Allogeneic Hematopoietic Cell Transplantation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RG1123691; NCI-2023-05599 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RG1123691 (Other: Fred Hutch/University of Washington Cancer Consortium); FHIRB0020155 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Acute Graft Versus Host Disease; Hematopoietic and Lymphatic System Neoplasm
MeSH Terms: interventions — Fecal Microbiota Transplantation; Parturition

STUDY DESIGN:
Intervention Model Description: The first 12 patients are assigned to the treatment group, remaining patients are randomized to treatment or placebo group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigators, treating physicians, staff, and subjects are blinded to study arm assignment (FMT vs. placebo).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (fecal microbiota transplant) (Experimental): Patients receive fecal microbiota capsules PO QD for 7 days
  Interventions: Drug: Fecal Microbiota Transplantation Capsule
- Group II (Placebo) (Placebo Comparator): Patients receive placebo PO QD for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fecal Microbiota Transplantation Capsule — Given PO
  Other Names: Fecal Microbiota Preparation Delivery Capsule; FMPCapDE; FMT Capsule DE; FMT Capsule Delivery; FMT DE Capsule
  Arms: Group I (fecal microbiota transplant)
Drug: Placebo — Given PO
  Arms: Group II (Placebo)

SUMMARY:
This randomized placebo-controlled double-blind phase II trial tests whether fecal microorganism (microbiota) transplantation prevents severe acute graft versus host disease in adults undergoing allogeneic hematopoietic cell transplantation (HCT). Fecal microbiota transplantation involves receiving processed fecal material orally after allogeneic HCT in order to establish a healthy gut microbiota. Gut microbiota undergoes major alterations during allogeneic HCT because of antibiotic exposures, nutritional changes, and chemotherapy administration. Establishing a healthy gut microbiota via fecal transplantation may help prevent acute graft versus host disease in patients undergoing allogeneic HCT.

DETAILED DESCRIPTION:
OUTLINE: The first 12 patients are assigned to group I, remaining patients are randomized to 1 of 2 groups.

GROUP I: Patients receive fecal microbiota capsules orally (PO) once daily (QD) for 7 days starting at the time of neutrophil engraftment and discontinuation of anti-bacterial antibiotics.

GROUP II: Patients receive placebo PO QD for 7 days starting at the time of neutrophil engraftment and discontinuation of anti-bacterial antibiotics.

After completion of study intervention, patients are followed up monthly until 12 months post-allogeneic HCT.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18
* Signed informed consent
* Able to take oral medications
* Planned T-replete allogeneic hematopoietic cell transplantation for any indication. History of prior transplantation is allowed
* Planned GVHD prophylaxis using one of the following regimens:

  * Calcineurin inhibitor (tacrolimus or cyclosporine) plus methotrexate
  * Calcineurin inhibitor (tacrolimus or cyclosporine) plus mycophenolate mofetil (MMF)
  * Sirolimus plus cyclosporine plus MMF
  * Post-transplant cyclophosphamide plus calcineurin inhibitor (with or without MMF or sirolimus)
* One of the following HCT donor types:

  * Human leukocyte antigen (HLA)-matched sibling donor
  * 9/10 or 10/10 HLA-matched unrelated donor
  * HLA- haploidentical donor
  * Cord blood
* Willing to use at least 1 accepted method of contraception until day 180 after transplant and agree to not donate eggs/sperm for 180 days after
* Not pregnant or breast feeding
* ELIGIBILITY CRITERIA FOR RANDOMIZATION: Absolute neutrophil count (ANC) recovery to > 0.5 x 10^9/L from nadir, without ongoing growth factor support
* ELIGIBILITY CRITERIA FOR RANDOMIZATION: Discontinuation of all antibacterial antibiotics (except those used for Pneumocystis jiroveci prophylaxis) for 2 days
* ELIGIBILITY CRITERIA FOR RANDOMIZATION: Resolution of all acute toxicities (other than anemia and thrombocytopenia) to Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or lower
* ELIGIBILITY CRITERIA FOR RANDOMIZATION: Ability to swallow capsules
* ELIGIBILITY CRITERIA FOR RANDOMIZATION: No grade II-IV acute GVHD
* ELIGIBILITY CRITERIA FOR RANDOMIZATION: No moderate to severe chronic GVHD
* ELIGIBILITY CRITERIA FOR RANDOMIZATION: No concurrent antibiotics to treat infections. Prophylactic antiviral and antifungal antibiotics used to prevent infections are allowed

Exclusion Criteria:

* Severe food allergy in the form of anaphylaxis or attributable symptoms requiring hospitalization
* History of chronic aspiration or conditions predisposing to aspiration (e.g. neuromuscular disorders)
* Receiving or planned to receive other experimental agents (including ex vivo T-cell depletion) to prevent GVHD. The use of other experimental agents is prohibited unless approved by the principal investigator (PI) of the other trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Grade III-IV acute graft versus host disease (GVHD) | Up to 6 months post hematopoietic cell transplantation (HCT)
  Based on International Blood and Marrow Transplantation Research (IBMTR) criteria and measured as a probability

SECONDARY OUTCOMES:
Grade II-IV acute GVHD | Up to 180 days post HCT
  Based on IBMTR criteria and measured as a probability
Non-relapse mortality | Up to 180 days post HCT
  Death not due to relapse/progression of the underlying hematologic disorder and measured as a probability
Clostridium difficile diarrhea | Up to 180 days post HCT
  Based on a positive stool assay in the consistent clinical setting (e.g. diarrhea) and measured as a probability
Chronic GVHD | At 12 months post-HCT
  Diagnosis based on the National Institutes of Health Consensus Criteria (PMID: 25529383)

CONTACTS AND LOCATIONS:
Overall Officials: Armin Rashidi, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reddi S, Senyshyn L, Ebadi M, Podlesny D, Minot SS, Gooley T, Kabage AJ, Hill GR, Lee SJ, Khoruts A, Rashidi A. Fecal microbiota transplantation to prevent acute graft-versus-host disease: pre-planned interim analysis of donor effect. Nat Commun. 2025 Jan 25;16(1):1034. doi: 10.1038/s41467-025-56375-y. PMID 39863610

DOCUMENTS (1):
  • Informed Consent Form (2025-09-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT06026371/ICF_000.pdf